CLINICAL TRIAL: NCT06938841
Title: Maintaining the Acute Therapeutic Effect of rTMS in Treatment-Resistant Depression (Maitr-De)
Brief Title: Maintenance rTMS for Depression (Maitr-De)
Acronym: Maitr-De
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Zafiris Daskalakis, MD, PhD., University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 811708
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder; Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Clustered maintenance rTMS (Experimental): Clustered maintenance treatment involves administering four sessions of rTMS over a two-day span, conducted once per month for six months.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS) - Clustered maintenance rTMS:
- Standard maintenance rTMS: (Active Comparator): Standard maintenance rTMS involves a course of rTMS with once-weekly sessions for 6 months.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS) - Standard maintenance rTMS:
- sham maintenance rTMS (Placebo Comparator): Somatosensory-matched placebo rTMS is delivered according to either standard or clustered maintenance schedules over a six-month period (50/50% allotment). Patient's maintenance protocol parameters will otherwise mirror those used during their acute treatment with identical cortical targets, stimulation intensity, frequency, and duration. Sham TMS-EEG will be conducted by rotating the coil 90 degrees while maintaining contact with the scalp. This standard practice prevents current induction while replicating the auditory click associated with TMS, ensuring comparable EEG recordings
  Interventions: Device: Transcranial Magnetic Stimulation (TMS) -- Sham maintenance rTMS

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) - Standard maintenance rTMS: — In this approach, patients who were treated with rTMS five days per week during their acute episode receive less frequent treatments during a taper period (for example treatment three days per week followed by two sessions per week) with a gradual transition into a maintenance schedule. For example, the maintenance schedule might begin with a single weekly session for one or two months and then the intensity is reduced to one session every two weeks (and possibly then one session every three or four weeks).
  Arms: Standard maintenance rTMS:
Device: Transcranial Magnetic Stimulation (TMS) - Clustered maintenance rTMS: — Clustered maintenance rTMS typically involves around 4 TMS sessions applied over 2 days, at 1-month intervals. Our team initially developed this approach based upon preclinical TMS studies (for example (Maeda et al. 2000)) suggesting that rTMS treatment effects may accumulate when applied over multiple sessions in a shorter period of time (Maeda et al. 2000).
  Arms: Clustered maintenance rTMS
Device: Transcranial Magnetic Stimulation (TMS) -- Sham maintenance rTMS — Sham treatment will be administered as either standard or clustered maintenance rTMS for 6 months period using a sham coil. The intervention target will be located via a Brainsight TMS Navigator (Brainsight, Montreal, Canada). For safety reasons, the individual TMS intensity will be limited to 130% of the individual resting motor threshold.
  Arms: sham maintenance rTMS

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) has emerged as a promising intervention for treatment-resistant depression (TRD), yet substantial uncertainties persist regarding its efficacy as a maintenance treatment. This prospective study seeks to investigate the efficacy of maintenance rTMS in individuals with TRD who have previously responded to an acute course of rTMS. In the R61 phase of the study, we will recruit 75 participants across three study sites, the University of California San Diego, Weill Cornell Medicine, and Australian National University, into a double-blind, three-arm maintenance treatment trial. In this trial, participants will be randomized to receive either standard maintenance rTMS, clustered maintenance rTMS, or sham maintenance rTMS for a duration of 6 months. Our primary aim is to examine the efficacy of maintenance rTMS on sustaining connectivity between the dorsolateral prefrontal cortex (DLPFC) and subgenual cingulate cortex (SGC) measured through concurrent TMS and electroencephalography (TMS-EEG) at baseline and every six weeks throughout the 6-month treatment period. We will also assess changes in depressive symptom severity using clinical scales, including the Montgomery-Asberg Depression Rating Scale (MADRS) as a secondary outcome measure. It is hypothesized that stimulation with clustered maintenance rTMS will demonstrate superiority in sustaining DLPFC-SGC connectivity compared with standard maintenance rTMS and sham maintenance rTMS

ELIGIBILITY:
Inclusion Criteria:

* 1. They met criteria for a DSM-5 diagnosis of a Major Depressive Episode (MDE) during the index episode of depression for which they have received an acute rTMS treatment course.

  2. Meet criteria for either response or remission from their initial depressive illness. The MINI assessment timeline will be adjusted to allow scoring of illness symptoms prior to rTMS response. Response to acute course of treatment is defined as either a MADRS score of <7, or a MADRS score of 7-19, plus evidence of having met response criteria on either the MADRS or another structured depression rating scale. The response is defined as a >50% reduction in the total score from the start to the end of treatment.

  3. Their initial rTMS treatment course must have consisted of at least 15 rTMS treatment sessions.

  4. People between the ages of 18 and 80 at the time of screening. A written statement from the referring physician will be required to confirm that the participant demonstrates the capacity to consent.

  5. Able to read, understand, and provide written, dated informed consent prior to screening. Proficiency in English sufficient to complete questionnaires / follow instructions during TMS-EEG assessments and iTBS interventions. Stated willingness to comply with all study procedures, including availability for the duration of the study, and to communicate with study personnel about adverse events and other clinically important information.

  6. In good general health, as evidenced by medical history. 7. Agreement to adhere to Lifestyle Considerations throughout study duration. 8. If a person of child-bearing potential is: must take a pregnancy test at the screening visit, with results confirmed as negative by study staff

Exclusion Criteria:

* 1. Pregnancy 2. History of or current psychotic disorder or depression with psychotic features 3. Severe borderline personality disorder based on clinical assessment. 4. Diagnosis of Intellectual Disability or Autism Spectrum Disorder 5. Current moderate or severe substance use disorder or demonstrating signs of acute substance withdrawal 6. Clinically significant suicidal ideation with plan 7. Any history of ECT (greater than 8 sessions) without a clinical meaningful response in the current episode.

  8. Recent (during the current depressive episode) or concurrent use of rapid-acting antidepressant agent (i.e., ketamine or a course of ECT) in the last 30 days 9. History of significant neurologic disease, including dementia, Parkinson's or Huntington's disease, brain tumor, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma 10. Untreated or insufficiently treated endocrine disorder. 11. Contraindications to receiving rTMS (e.g., metal in head, history of seizure, known brain lesion) 12. Treatment with an investigational drug or other intervention within the study period 13. Unstable symptoms between screening and baseline as defined by a ≥ 30% change in MADRS score.

  14. Require a benzodiazepine with a dose > lorazepam 2 mg/day or equivalent or any anticonvulsant (with the exception of Gabapentin).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Aim: To evaluate the effects of two active rTMS maintenance treatments (i.e., standard and clustered) compared to sham maintenance rTMS on DLPFC-SGC connectivity. | 6-months
  Our primary aim is to examine the efficacy of maintenance rTMS on sustaining connectivity between the dorsolateral prefrontal cortex (DLPFC) and subgenual cingulate cortex (SGC) measured through concurrent TMS and electroencephalography (TMS-EEG) at baseline and every six weeks throughout the 6-month treatment period

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - University of California, San Diego, San Diego, California
  - Weill Cornell Medicine, New York, New York
- Australian National University, Canberra, Australian Capital Territory, Australia

IPD SHARING:
Plan to Share IPD: No